CLINICAL TRIAL: NCT00156403
Title: Hereditary Pancreatitis Amlodipine Trial(H-PAT): A Pilot Study
Brief Title: A Pilot Study of Use of Calcium Channel Blocker to Decrease Inflammation and Pain in Hereditary Pancreatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0505070; CReFF Award, GCRC U Pittsburgh; National Pancreas Foundation
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-12-17 (Estimated); Status verified 2007-12

CONDITIONS: Pancreatitis
Keywords: pancreatitis, hereditary; trypsinogen, cationic; pilot study
MeSH Terms: conditions — Pancreatitis; Hereditary pancreatitis | interventions — Amlodipine; Pharmaceutical Preparations

INTERVENTIONS:
Drug: amlodipine (drug)

SUMMARY:
This pilot study is a feasibility, safety, and preliminary benefits study to look at whether giving the calcium channel blocker amlodipine to people with hereditary pancreatitis as a prophylactic measure can reduce the inflammatory process in the pancreas.

DETAILED DESCRIPTION:
Hereditary Pancreatitis is a rare, autosomal dominantly inherited condition causing mutations in the cationic trypsinogen gene. These mutations lead to excessive activation of trypsinogen within the pancreatic acinar cells and subsequent pancreatic inflammation. Clinically, this may be observed as recurrent acute pancreatitis, chronic pancreatitis, and eventual complications of exocrine and endocrine pancreatic insufficiencies and pancreatic adenocarcinoma. Currently, there are no specific treatment or prophylactic measures for this condition.

Calcium is the physiologic switch to activate trypsinogen. It has recently been found that the mutation sites affect how tightly calcium binds to trypsinogen, with mutations leading to excessive calcium binding and subsequent excessive trypsinogen activation. This study is to obtain baseline data on whether the prophylactic use of a long-acting calcium channel blocker, amlodipine, would lead to decrease in the inappropriate activation of trypsinogen, and thereby decrease the subsequent pancreatic inflammation.

Up to 15 subjects, aged 6 years and above, with mutations in the cationic trypsinogen gene (PRSS1) will be recruited and undergo a 16-week trial. This will include a one-month baseline symptoms assessment (daily symptoms diary) and blood pressure measurements (with an automated home blood pressure monitor). Subsequently, subjects will be placed on between 2.5 - 10 mg amlodipine po qd (with a weaning up and weaning down phase) for approximately 10 weeks. They will continue to fill out daily symptoms diary, blood pressure measurements (to ensure there are no decreases), fill out periodic quality of life questionnaires, and undergo periodic blood testing for routine biochemistry as well as more specialized testing for proteomics and other inflammatory cytokines analysis.

The study has three main purposes: to determine whether the use of amlodipine appears to be safe in this patient population, to determine how frequently and how best to follow subjects while they are taking the medication, and to determine whether there are any indications of potential benefits to the medication (whether by decreased symptoms frequency/ severity or by inflammatory cytokines analysis).

A subsequent larger study would be designed based on the above results.

ELIGIBILITY:
Inclusion Criteria:

* mutation in cationic trypsinogen (PRSS1)gene
* age 6 years and above
* able to comply with study terms: taking daily oral medication, taking daily blood pressure, filling in daily symptoms diary, coming to all follow-up visits
* having some symptoms of pain from pancreas

Exclusion Criteria:

* combination of mutations in the 2 other loci associated with pancreatitis: Cystic fibrosis transmembrane regulator and serine protease inhibitor Kazal type 1 (having mutations in both genes)
* pancreatic insufficiency (exocrine and endocrine)
* already being on an antihypertensive medication
* contraindication to taking amlodipine (allergic reaction, severe renal failure (creatinine > 3 mg/dL; hepatic dysfunction signified by INR > 1.5)
* pregnancy or breastfeeding
* systemic disease that the investigators feel would place patient at undue risk of being placed on amlodipine
* newly-started (within past 3 months) pancreatic enzymes, acid blocking medication, antioxidants, or oral contraceptive medication

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8
Dates: Start 2005-08; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
safety of amlodipine: side effects, biochemistry, BP
efficacy: symptoms diary, SF-36, cytokines analysis

SECONDARY OUTCOMES:
feasibility: ease of obtaining patient symptoms information, whether subjects need to be followed up as frequently as designated in this pilot, whether doing regular laboratory tests changed management in any way (i.e. whether it was necessary)

CONTACTS AND LOCATIONS:
Overall Officials: David C Whitcomb, MD, PhD, Study Director — Chief, Division of Gastroenterology, Hepatology and Nutrition, University of Pittsburgh and University of Pittsburgh Medical Center, M2, C-Wing, Presbyterian Hospital, 200 Lothrop Street, Pittsburgh PA 15213
Locations (1):
- General Clinical Research Center, University of Pittsburgh, Pittsburgh, Pennsylvania, United States